CLINICAL TRIAL: NCT03942770
Title: Remote Alcohol Monitoring to Facilitate Abstinence Reinforcement With an Underserved Population
Brief Title: Remote Alcohol Monitoring to Facilitate Abstinence From Alcohol: Exp 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mikhail N Koffarnus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Mikhail N Koffarnus, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-324; R01AA026605 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Active Comparator: Group A (Intensive incentives) (Active Comparator): Group A will have the opportunity to earn payments based on the results of their breathalyzer screens. Participants will receive a compliance incentive per submitted sample regardless of the results, but will also have the opportunity to earn more incentives for providing negative results. For the first 3 weeks, these additional incentives will scale based on the number of consecutive days of sustained negative samples. For the remaining weeks incentives will be based on a randomized "prize" drawing.
  Interventions: Behavioral: Contingency Management
- Active Comparator: Group B (Prize-based incentives) (Active Comparator): Group B will have the opportunity to earn payments based on the results of their breathalyzer screens. Participants will receive a compliance incentive per submitted sample regardless of the results, but will only have the opportunity to earn more incentives based on a randomized "prize" drawing if they submit a negative sample.
  Interventions: Behavioral: Contingency Management
- Sham Comparator: Group C (Intensive incentives) (Sham Comparator): Group C serves as a direct control group to Group A and will follow the same incentive procedures, however participants will receive incentives regardless of the results of their samples.
  Interventions: Behavioral: Contingency management
- Sham Comparator: Group D (Price-based incentives) (Sham Comparator): Group D serves as a direct control group to Group B and will follow the same incentive procedures, however participants will receive incentives regardless of the results of their samples.
  Interventions: Behavioral: Contingency management
- No Intervention: Group E (no incentives) (No Intervention): Group E will have no monitoring intervention, they will only complete assessment sessions.

INTERVENTIONS:
Behavioral: Contingency Management — Monetary incentives are delivered to participants contingent upon on-time breathalyzer submissions and verified abstinence from alcohol.
  Other Names: Contingent incentives
  Arms: Active Comparator: Group A (Intensive incentives); Active Comparator: Group B (Prize-based incentives)
Behavioral: Contingency management — Monetary incentives are delivered to participants contingent upon on-time breathalyzer submissions only with no contingency on alcohol use.
  Other Names: Noncontingent incentives
  Arms: Sham Comparator: Group C (Intensive incentives); Sham Comparator: Group D (Price-based incentives)

SUMMARY:
Directly reinforcing abstinence from alcohol with monetary incentives is an effective treatment for alcohol dependence, but barriers in obtaining frequent, verified biochemical measures of abstinence limit the dissemination of this treatment approach. As our feasibility study demonstrates, remote breathalyzer monitoring drastically improves the practicality of delivering an alcohol contingency management intervention. In Experiment 2, we will test whether the addition of remote abstinence incentives to treatment as usual improves outpatient treatment outcomes and prevents relapse following inpatient detoxification at a regional hospital system. We will also assess whether readmission rates are reduced using a newly developed smartphone app and breathalyzer.

ELIGIBILITY:
Inclusion Criteria:

* Recently completed or currently completing an alcohol detoxification program through the Carilion Clinic or University of Kentucky Healthcare system.
* Meet DSM-V criteria for alcohol use disorder.
* Abstinent from alcohol at the time of consent.

Exclusion Criteria:

* Alcohol use disorder is secondary to another substance use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pattern of abstinence from alcohol during intervention | up to 66 weeks
  Breathalyzer assessments will be collected during the treatment period. This outcome measure will consist of the percentage of days without alcohol use as detected by the breathalyzers.
Treatment acceptability | A total of 12 assessment sessions spanning over a 66 week period
  Participant ratings of treatment acceptability on a customized Treatment Acceptability questionnaire will be collected during assessment sessions. Each question will be scored from 1 (low) to 4 (high) and will assess distinct components of the treatment. Questions will be interpreted and scored individually and not be summed together.
Time to relapse | A total of 12 assessment sessions spanning over a 66 week period
  For this outcome, we will conduct survival analyses to compare relapse across study groups.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky Healthcare, Lexington, Kentucky
  - Virginia Tech Carilion, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Final research data for this project will be made as available as possible, while safeguarding the privacy of participants and protecting all confidential and proprietary data. Data will be available for use after the main findings from the final dataset have been accepted for publication. The data and associated documentation will only be made available to users under a Data Use Agreement that provides for 1) a commitment to using the data only for research purposes and not to identify any individual participant and 2) a commitment to destroying or returning the data after analyses are completed. To ensure compliance with HIPAA regulations, only a Limited Data Set will be available for use. The method of data release will be determined on a case-by-case basis depending upon the amount and type of data required.
Supporting Information: Study Protocol, SAP, ICF